CLINICAL TRIAL: NCT01466231
Title: Phase II Study of Everolimus in Refractory Testicular Germ Cell Cancer.
Brief Title: Everolimus in Refractory Testicular Germ Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Slovakia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCTSK002
Record Dates: First submitted 2011-10-31; First posted 2011-11-07 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Germ Cell Tumor
Keywords: refractory germ cell cancer; everolimus
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- everolimus 10 mg po daily (Experimental): everolimus 10 mg po daily
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Tablets p.o. 10 mg daily until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements.
  Other Names: Afinitor

SUMMARY:
Everolimus in refractory testicular germ cell cancer. Everolimus 10 mg /day/ is administered to the patient until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements. Feasibility of surgical resection will be assessed after every 2 cycles of the treatment in patients with partial response.

DETAILED DESCRIPTION:
Treatment Schedule: Everolimus will be administered at a dose of 10mg/day orally once a day. One cycle of therapy consists of 28 days.

Estimated duration of treatment: Until progression, unacceptable toxicity, complete response or inability of the subject to comply with study requirements.

Feasibility of surgical resection will be assessed after every 2 cycles of the treatment in patients with partial response.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Men aged 18 years or older
3. ECOG performance status: 0-2,
4. Histological confirmed extracranial primary germ cell cancer, seminoma, or nonseminoma
5. Rising serum markers (i.e., alpha-fetoprotein and human chorionic gonadotropin) on sequential measurement or biopsy-proven unresectable germ cell cancer
6. Refractory GCTs e.g. patients relapsing after high-dose chemotherapy or for patients non fit enough for high-dose chemotherapy
7. Primary mediastinal GCTs in first relapse
8. Patient's disease must not be amenable to cure with either surgery or chemotherapy in the opinion of investigator,
9. Measurable disease radiological
10. Adequate hematologic function defined by WBC > 4000/mm3, platelet count > 100 000/mm3 and hemoglobin level > 9g/dl.
11. Adequate liver function defined by a total bilirubin level < 1.5 ULN, and ALT, AST < 2,5 ULN and adequate renal function defined by serum creatinine ≤ 1.5 x ULN.
12. At least 2 weeks must have elapsed since the last radiotherapy and/or chemotherapy before study entry,
13. At least 4 weeks must have elapsed since the last major surgery
14. Complete recovery from prior surgery, and/or reduction of all adverse events from previous systemic therapy or radiotherapy to grade 1,
15. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, -

Exclusion Criteria:

1. Patients who do not fit inclusion criteria,
2. Other prior malignancy except successfully treated non melanoma skin cancer
3. Prior treatment with mTOR inhibitor
4. No other concurrent approved or investigational anticancer treatment, including surgery, radiotherapy, chemotherapy, biologic-response modifiers, hormone therapy, or immunotherapy
5. Female patients,
6. Patients infected by the Human Immunodeficiency Virus (HIV),
7. Patients with other severe acute or chronic medical condition, or laboratory abnormality that would impair, in the judgment of investigator, excess risk associated with study treatment, or which, in judgment of the investigator, would make the patient inappropriate for entry into this study,
8. Inability of oral intake, or drug absorption (e.g. malabsorption syndrome)
9. Hypersensitivity to any compound of the drug,
10. Sexually active men not using effective birth control if their partners are women of child-bearing potential.
11. Patients with active CNS metastasis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Response rate | 36 month
  according RECIST criteria version 1.1

SECONDARY OUTCOMES:
Favorable response rate | 36 month
  complete response with chemotherapy and/or surgery, partial response marker negative.
Clinical benefit rate | 36 month
  (complete and partial response and stable disease > 6 months)
Progression-free survival | 36 month
  expressed as median and as 12-weeks post-treatment initiation continuous progression-free survival rate
Toxicity | 36 month
Frequency of grade III and IV adverse events | 36 month
Association between clinical outcome and biomarkers | 36 month
Serum tumor markers response | 36 month
  >90% decline of AFP and/or HCG

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Mardiak, Prof, Principal Investigator — National Cancer Institute (NCI); Michal Mego, Ass.prof., Study Chair — National Cancer Institute, Slovakia
Locations (1):
- National Cancer Institute, Bratislava, Slovakia